CLINICAL TRIAL: NCT04159857
Title: Efficacy and Safety Comparison of an Innovative Two-hand vs. Conventional One-hand Technique for Fetal Head Manual Extraction During a Low Transverse Cesarean Section: A Randomized Controlled Study
Brief Title: Hand Forceps vs. Conventional One-hand Technique for Fetal Head Extraction During Cesarean Section
Acronym: Hand forceps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Reading Hospital and Medical Center (Other)
Responsible Party: Principal Investigator, Xuezhi (Daniel) Jiang, MD, Research and Clerkship Director of OBGYN, The Reading Hospital and Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB 028-18
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy Related; Delivery Complication; Cesarean Delivery Affecting Fetus
Keywords: hand forceps, cesarean section, one-hand technique, two-hand technique, fetal head extraction

STUDY DESIGN:
Intervention Model Description: Arm 1: Fetal head is extracted by conventional one-hand (in hysterotomy) technique during the C-section Arm 2: Fetal head is extracted by an innovative two-hand (in hysterotomy) technique during the C-section
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-hand (Active Comparator): During LTCS, the fetal head traditionally is delivered by one-hand manual extraction (a surgeon inserts one hand into the uterus via the hysterotomy and lifts the fetal head out of maternal pelvis, subsequently significant abdominal pressure is required to squeeze the fetal head out of hysterotomy) along with application of significant abdominal/fundal pressure.
  Interventions: Procedure: Fetal head extraction technique during the cesarean section
- Two-hand (Experimental): An innovative approach to manual head extraction, with surgeon's both hands formed as a pair of forceps, has been used by the PI of this study for years during the LTCS for head extraction in the difficult situations described above without complication, often time it was used after one hand approach failed to deliver the infant, vacuum/forceps and abdominal pressure usually was not needed in these cases.
  Interventions: Procedure: Fetal head extraction technique during the cesarean section

INTERVENTIONS:
Procedure: Fetal head extraction technique during the cesarean section — see above for the description about one-hand and two-hand fetal head extraction technique

SUMMARY:
The aim of the study is to assess the efficacy and safety of an innovative two-hand (hand forceps) fetal head extraction technique during the transverse cesarean sections (LTCS) by comparing with the conventional one-hand technique used worldwide for centuries.

The primary research question of the study is whether two-hand fetal head extraction technique results in quicker head delivery. The secondary research question is whether two-hand technique would cause increased incidence of extension of uterine incision as well as other adverse events while compared to conventional one-hand technique.

Our hypothesis is that two-hand technique would speed up fetal head delivery without increasing the risk of extension of uterine incision as well as other adverse events, in the meantime, maternal discomfort will be significantly reduced since fundal pressure will not be required during the fetal head delivery.

DETAILED DESCRIPTION:
It is not unusual that obstetricians struggle with head delivery during the LTCS, when it occurs, it can not only lead to substantial personal distress for the individual surgeons, but also frequently require operative delivery (vacuum or forceps), deliberate extension of hysterotomy (i.e. inverted T-incision on the uterus), or partial transection of rectus muscles which may be associated with higher maternal and neonatal morbidity as well as obstetrical and surgical complications for the future pregnancy.

During LTCS, the fetal head traditionally is delivered by one-hand manual extraction (a surgeon inserts one hand into the uterus via the hysterotomy and lifts the fetal head out of maternal pelvis, subsequently significant abdominal pressure is required to squeeze the fetal head out of hysterotomy) along with application of significant abdominal/fundal pressure. While abdominal pressure may cause maternal discomfort, in some cases (i.e. obesity with big pannus or thickened anterior abdominal wall, high-floating/mobile fetal head above the hysterotomy incision, tight rectus muscles, tight U- or V-shaped transverse hysterotomy incisions, deflexed fetal head), application of vacuum or obstetrics forceps, deliberate extension of hysterotomy incision either transversely or vertically (inverted t-incision), excessive uterine fundal pressure or partially transection of rectus abdominis muscles may be required. In addition to maternal discomfort due to increased fundal pressure, the result often is either traumatic or undue delay in delivering the infant. An innovative approach to manual head extraction, with surgeon's both hands formed as a pair of forceps, has been used by the PI of this study for years during the LTCS for head extraction in the difficult situations described above without complication, often time it was used after one hand approach failed to deliver the infant, vacuum/forceps and abdominal pressure has never been needed in these cases. One potential argument against two-hand technique is that it could increase the risk of extension of uterine incision since two hands require more intrauterine space than one hand. This was never the case based on PI's personal experience, however, no evidence-based data is available to support or recommend against the clinic use of this two-hand approach. This study was designed to compare the efficacy and safety outcome of two different head extraction techniques in a randomized controlled study. If two-hand approach was approved to be a safe and more effective way for fetal head extraction during LTCS, it would potentially reduce the likelihood of application of vacuum/forceps and deliberate extension of hysterotomy (i.e. Inverted T-incision which may disqualify the patient for trial of labor after C-section [TOLAC] for the future pregnancy since the risk of uterine rupture may be significantly increased after t-incision was made in the previous pregnancy), in addition to significant mental stress reduction for surgical team and relief of maternal discomfort caused by excessive fundal pressure.

This study consists of two phases with phase 1 being a prospective case series study for safety data collection, and phase 2 being a randomized control study that includes two study groups (two-hand vs. one-hand).

Phase 1: all OBGYN residents will be trained to learn and grasp the two-hand technique via watching educational videos and practicing in simulation lab. The technique includes two key steps. Step 1, insert one hand into the hysterotomy to assess position of fetal head with vast majority of cases being occiput transverse, then insert the second hand to form a hand-forceps to cover both ears and lower jawbones on the side. Surgeon's fingers need to pass mandibles to secure sufficient grip to prevent slipping. Step 2, pulling fetal head out of hysterectomy, Step 3, delivering posterior shoulder followed by anterior shoulder once fetal head was delivered. Residents must be signed off by PI based on above criteria prior to administering the two-hand technique in real patients. Residents will be allowed to apply two-hand technique when they encounter difficulty delivering fetal head by one-hand technique and prior to applying vacuum or forceps assisted delivery or extending the hysterotomy (inverted T incision). Phase 1 will primarily focus on safety assessment of two-hand technique, therefore, data on extension of uterine incision and neonatal outcome will be collected. Consent will not be required for the phase 1 since hand-forceps technique will only be used after conventional one-hand technique failed and before more invasive vacuum or metal forceps is applied. If increase in negative neonatal outcome is not noted and none of negative outcomes was considered being associated with two-handed technique, after 30 cases were assessed, investigators will move on to phase 2 after informing RAC and IRB. Incidence of spontaneous extension of uterine incision will not be considered primary end point for the phase 1 since extension can be attributed to many factors (i.e. thin lower uterine segment due to prolonged labors, bending the hand while lifting fetal head out of lower pelvis, etc.) rather than the two-hand technique, and it will be unlikely to distinguish the real cause of extension in phase 1 without doing a head-to-head comparison. The incidence of one handed technique leading to extended hysterotomy (background incidence) is unknown thus it will be unrealistic to compare the incidence of extension of hysterotomy observed in phase 1 with background incidence either.

Phase 2: After informed consent was obtained either in the women's health center (WHC) or labor & delivery (L&D), study subjects will be recruited for undergoing an elective cesarean section. Inclusion criteria include gestational age 37 weeks or above with cephalic presentation, planned low transverse uterine incision, cervical dilation <= 6cm, station < 0. All recruited subjects will be randomized to the study or control arm in L&D according to a computer generated randomized schedule. Group assignment will be concealed in an envelope labeled with subject number and opened prior to C-section. All deliveries will be timed by a designated staff using stopwatches from the time of entry into the uterus (insertion of a surgeon's hand into uterus through the fully transected lower uterine segment) until the full delivery of the fetal head. Cesarean section will be timed by OR staff as a matter of routine. Although it may be easy to learn and grasp the skill of two-hand technique, all house staffs must be trained to use both hands for head extraction in phase 1. If delivery was not imminent after attempting at manual extraction with one-hand technique in control group, then the surgeon should proceed with two-hand technique prior to extending the hysterotomy incision and/or applying vacuum or forceps, and vice versa. The study will be registered with clinicaltrials.gov. The number of patients approached for study, met criteria, recruited, and withdrawal will be tracked and recorded. Both intention-to-treat and per-protocol analyses will be conducted. Aside from an electronic medical record (EPIC), additional information will be recorded in a separate datasheet such as time from entry of uterus to delivery of fetal head (U-D interval), whether excessive fundal pressure was applied (defined as a pressure that was applied by both surgeons or one of surgeons standing with both feet in a tiptoe position and keeping both arms and elbows straight so that shoulders are directly over surgeon's hands), whether initial planned technique fails and the alternative technique succeeds, any laceration or extension of hysterotomy incision (whether C-section is elective or not, cervical dilatation and station prior to C-section, thickness of subcutaneous tissue (>6 cm or <=6 cm), head engaged or high floating, direction [horizontal, vertical, oblique] and location[apex of hysterotomy incision, inferior aspect of hysterotomy incision, cervical laceration]) of extension, whether deliberate extension of hysterotomy incision was made and location(lateral extension, inverted T-incision), whether vacuum or forceps was applied. Time from entry of uterus and fetal head delivery as a primary outcome as well as other continuous variables with normal distribution, such as age, maternal weight and BMI, will be analyzed using student's t-test. Non-parametric methods will be applied to ordinal data or non-normally distributed continuous data. Categorical variables (i.e. success rate of initial attempt at per-protocol extraction technique) will be analyzed using Chi-square test. SPSS or SAS will be used for statistical analysis. P<0.05 is deemed statistically significant.

Mean U-D intervals using one-hand technique for manual extraction range from 30-60 seconds in the literature (1-5). Investigators used 45+/-15 seconds as a mean U-D interval, one sided test, α level of 0.05, 80 % power to detect 30% reduction in U-D interval, a total sample size of 42 (21 for each group) will be needed. If 20% of study withdrawal was taken into account, a total of 52 patients need to be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) 37 weeks or above with cephalic presentation
* Planned low transverse uterine incision
* Cervical dilation <= 6cm
* Station < 0.

Exclusion Criteria:

* Preterm GA <37 weeks
* Planned classical C-section
* Unable or unwilling to afford abdominal pressure during the delivery of fetal head
* Advanced cervical dilation >6cm
* Station >=0

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-01-28 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Time needed for fetal head delivery | 2 year
  Time from entry of uterus to delivery of fetal head (U-D interval)

SECONDARY OUTCOMES:
Extension of hysterotomy | 2 year
  incidence of extension of uterine incision as well as other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xuezhi (Daniel) Jiang, MD, Principal Investigator — Reading Hospital of Tower Health
Locations (1):
- Reading Hospital Labor & Delivery, West Reading, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arad I, Linder N, Bercovici B. Vacuum extraction at cesarean section--neonatal outcome. J Perinat Med. 1986;14(2):137-40. doi: 10.1515/jpme.1986.14.2.137. PMID 3735047